CLINICAL TRIAL: NCT04271072
Title: The Role of Cerebrospinal Fluid and Serum Inflammatory Biomarkers in Predicting Perinatal Depression and Persistent Pain After Cesarean Delivery
Brief Title: CSF/Serum Biomarkers in Predicting PND/Persistent Pain After Cesarean
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104111
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Perinatal Depression; Chronic Pain
Keywords: Neuroinflammation; Biomarker; Cesarean delivery; Cytokines; Cerebrospinal fluid
MeSH Terms: conditions — Chronic Pain; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and CSF samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Parturients that underwent cesarean delivery and is POSITIVE for the composite outcome of either:
  * perinatal depression (Edinburgh postnatal depression scale >=10 during pregnancy or within 3 months after delivery), and/or
  * persistent pain (pain score >=3 at pelvic or lower abdominal areas at 3 months after delivery)
  Interventions: Other: No intervention
- Control: Parturients that underwent cesarean delivery and is NEGATIVE for the composite outcome of both:
  * perinatal depression (Edinburgh postnatal depression scale >=10 during pregnancy or within 3 months after delivery), AND
  * persistent pain (pain score >=3 at pelvic or lower abdominal areas at 3 months after delivery)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim is to investigate if inflammatory biomarkers in the blood and cerebrospinal fluid (CSF) are associated with the development of perinatal depression and/or persistent pain after cesarean delivery.

This study will obtain CSF and blood samples in 70 parturients. All parturients will be assessed for perinatal depression and persistent pain, and the presence/absence of these outcomes will be correlated to changes in the inflammatory biomarkers within the samples collected. If present, consistent changes in biomarkers correlating with perinatal depression or persistent pain may be utilised as a predictive tool and facilitate early treatment for these conditions.

DETAILED DESCRIPTION:
Persistent pain and perinatal depression (PND) contribute significantly to maternal morbidity and mortality after cesarean delivery. Neuroinflammation has been associated with both persistent pain and perinatal depression, and may therefore be a common etiological process, however, little is known of the association between neuroinflammation and persistent pain or PND in parturients undergoing cesarean delivery.

Aim 1: To compare neuroinflammatory cytokine profiles (in CSF and plasma samples within 48 hours after surgery) between the cohort of parturients that develop the composite outcome of persistent pain or PND (defined below), versus the cohort of parturients that did not develop this outcome.

Aim 2. To determine the correlation between the neuroinflammatory cytokine profiles of CSF and plasma.

Exploratory aim: To determine the change in plasma inflammatory cytokine profile from the antenatal to the postnatal period, and correlate this change with preoperative quantitative sensory tests, acute postsurgical pain severity, and development of persistent pain and/or PND. To examine proteomics in CSF and correlate with persistent pain and/or PND.

This is a prospective cohort study of 70 adult parturients undergoing elective cesarean delivery at Duke University Hospital. After obtaining informed consent, baseline demographic data, the Edinburgh Postnatal Depression Scale (EPDS), mechanical temporal summation (MTS), and pain-pressure threshold (PPT) tests will be administered. During IV cannulation, 10ml of blood will be collected, and up to 10ml CSF will be collected during spinal anesthesia. After cesarean delivery, pain scores, analgesia requirements, and data on adverse events will be collected. Additional 10ml of blood will be collected within 48 hours post-surgery during inpatient hospital stay. During the routine 6-week postnatal follow up, EPDS scores will be recorded, and at 3-months, EPDS and persistent pain assessment will be conducted over the phone.

Based on a composite endpoint of persistent pain (pain at 3 months after surgery) or PND (EPDS of 10 or greater, during pregnancy or within 3 months after delivery), parturients will be stratified into "study" or "control" cohorts. Using a validated multiplex quantitative proteomic approach, candidate biomarkers will be quantified and correlated against the composite outcome using two-sided Mann-Whitney U test. Correlation between CSF and plasma cytokines will be assessed using spearman correlation. The exploratory aim will be analyzed with generalized linear models.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class 2 and 3
* English speaking
* 18 years or older
* Singleton pregnancy
* Gestational age > 37 weeks
* Scheduled cesarean delivery under spinal or combined spinal epidural anesthesia

Exclusion Criteria:

* Intravenous drug or chronic opioid use
* Anti-depressant or anxiolytic drug use
* Allergy to standard of care drugs
* Cesarean delivery under general anesthesia or epidural anesthesia
* Pre-eclampsia needing magnesium sulfate
* Chronic PO/IV analgesic or glucocorticoids
* History of chronic pain syndromes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant parturients are eligible
Study Population: Tertiary care hospital, specialist obstetric unit
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Perinatal depression | Up to 3 months after delivery
  Edinburgh postnatal depression scale >=10 (minimum 0, maximum 30, increasing score indicates higher likelihood of depression)
Persistent pain: Pain score | Up to 3 months after delivery
  Pain score >=3 at pelvic or lower abdominal areas (minimum 0, maximum 10, higher score indicates greater pain)
Inflammatory cytokines/biomarkers | Up to 24 hours after surgery
  Biomarkers from CSF and plasma samples will be quantified using Meso Scale Discovery multiplex kit (K15210D), for:
  CRP, Eotaxin, Eotaxin-3, FGF (basic), ICAM-1, IFN-γ, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12/IL-23p40, IL-13, IL-15, IL-16, IL-17A, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, PlGF, SAA, TARC, Tie-2, TNF-α, TNF-β, VCAM-1, VEGF-A, VEGF-C, VEGF-D, VEGFR-1/Flt-1.
  The levels of these biomarkers will be compared between the group with depression/persistent pain, versus the group without depression/persistent pain.

SECONDARY OUTCOMES:
CSF compared to plasma inflammatory cytokines/biomarkers | Preoperative samples
  Biomarkers will be quantified using Meso Scale Discovery multiplex kit (K15210D), for:
  CRP, Eotaxin, Eotaxin-3, FGF (basic), ICAM-1, IFN-γ, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12/IL-23p40, IL-13, IL-15, IL-16, IL-17A, IP-10, MCP-1, MCP-4, MDC, MIP-1α, MIP-1β, PlGF, SAA, TARC, Tie-2, TNF-α, TNF-β, VCAM-1, VEGF-A, VEGF-C, VEGF-D, VEGFR-1/Flt-1
  The CSF and plasma levels of these biomarkers will be compared within each group (group with depression/persistent pain, versus group without depression/persistent pain)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Yurashevich, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohler CA, Freitas TH, Maes M, de Andrade NQ, Liu CS, Fernandes BS, Stubbs B, Solmi M, Veronese N, Herrmann N, Raison CL, Miller BJ, Lanctot KL, Carvalho AF. Peripheral cytokine and chemokine alterations in depression: a meta-analysis of 82 studies. Acta Psychiatr Scand. 2017 May;135(5):373-387. doi: 10.1111/acps.12698. Epub 2017 Jan 25. PMID 28122130
- [Background] Miller ES, Sakowicz A, Roy A, Yang A, Sullivan JT, Grobman WA, Wisner KL. Plasma and cerebrospinal fluid inflammatory cytokines in perinatal depression. Am J Obstet Gynecol. 2019 Mar;220(3):271.e1-271.e10. doi: 10.1016/j.ajog.2018.12.015. Epub 2018 Dec 14. PMID 30557551
- [Background] Osborne LM, Monk C. Perinatal depression--the fourth inflammatory morbidity of pregnancy?: Theory and literature review. Psychoneuroendocrinology. 2013 Oct;38(10):1929-52. doi: 10.1016/j.psyneuen.2013.03.019. Epub 2013 Apr 20. PMID 23608136
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Ji RR, Nackley A, Huh Y, Terrando N, Maixner W. Neuroinflammation and Central Sensitization in Chronic and Widespread Pain. Anesthesiology. 2018 Aug;129(2):343-366. doi: 10.1097/ALN.0000000000002130. PMID 29462012
- [Derived] Yurashevich M, Cooter Wright M, Sims SC, Tan HS, Berger M, Ji RR, Habib AS. Inflammatory changes in the plasma and cerebrospinal fluid of patients with persistent pain and postpartum depression after elective Cesarean delivery: an exploratory prospective cohort study. Can J Anaesth. 2023 Dec;70(12):1917-1927. doi: 10.1007/s12630-023-02603-2. Epub 2023 Nov 6. PMID 37932648